CLINICAL TRIAL: NCT06016452
Title: A Prospective Phase 2 Study of Chlorophyllin for the Management of Brain Radionecrosis in Patients With Diffuse Glioma
Brief Title: A Study of Chlorophyllin for the Management of Brain Radio-necrosis in Patients With Diffuse Glioma
Acronym: CHROME
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Collaborators: Bhabha Atomic Research Centre (BARC) (Unknown)
Responsible Party: Principal Investigator, Dr Archya Dasgupta, Assistant Professor, Radiation Oncology, Tata Memorial Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 900970
Record Dates: First submitted 2023-08-10; First posted 2023-08-29 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Diffuse Glioma; Radionecrosis of Brain; High Grade Glioma; Glioblastoma Multiforme
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — chlorophyllin

STUDY DESIGN:
Intervention Model Description: The proposed phase II prospective study will be split into two strata: Stratum A (symptomatic RN) and Stratum B (asymptomatic RN).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stratum A (Symptomatic) (Experimental): Response rates at 1 month with a combination of steroids and CHL in this study is expected to be 65% as compared to the standard 50% response with the use of dexamethasone alone. For the study with an α of 0.1 and power of 80%,50 pts will be needed to achieve the desired output. In the first stage, 22 patients will be needed for assessment and continued to stage 2 if >10 responses are seen.The stage 2 of the study will be considered successful if >29 responses are achieved using the pre-specified response assessment criteria.Considering an attrition rate of 10% from lack of follow-up and another 10% for disease progression, an estimated 60 patients will be accrued in stratum A with the purpose of achieving 50 patients with endpoints available for analysis.
  Interventions: Drug: Chlorophyllin
- Stratum B (Asymptomatic) (Experimental): This stratum includes pts without neurological worsening during imaging diagnosis of RN (asymptomatic RN).Approx 30% of patients continue to be neurologically/ radiologically stable or regression of imaging findings without need for further interventions (including corticosteroids).In the proposed study with the use of CHL, 45% patients are assumed to remain clinically and neurologically stable. With an α of 0.1 and power of 80%, 48 patients will be needed to achieve the desired outcome. In the first stage, 23 patients will be needed for assessment and continue to stage 2 if >6 responses are seen.
  The phase 2 study will be considered successful if >18 responses are achieved using the pre-specified response assessment criteria. Further considering an attrition rate of 10% from lack of follow-up and another 10% for disease progression, an estimated 58 patients will be accrued in stratum B with the purpose of achieving 48 patients with endpoints available for analysis.
  Interventions: Drug: Chlorophyllin

INTERVENTIONS:
Drug: Chlorophyllin — Chlorophyllin is a water-soluble compound obtained from the green plant pigment called chlorophyll. It has been shown to have anti-cancer, anti-bacterial, anti-viral, anti-inflammatory, and antioxidant properties. It is also used as an oral formulation and is an over-the-counter drug in various countries, and also as a food coloring agent.
  Other Names: Stratum A (Symptomatic); Stratum A (Asymptomatic)

SUMMARY:
Diffuse gliomas are common tumors involving the brain. They are usually treated by surgery followed by radiation and chemotherapy. Radiotherapy is used for the treatment of brain tumors which causes damage to the tumor cells. However, radiotherapy can also affect the surrounding healthy cells in the brain, causing inflammation and swelling in the region, which is known as radio necrosis (RN). This is considered a late side effect of radiation and is seen in 10-25% of patients treated with radiation for brain tumors. Sometimes, radionecrosis can be detected on routine imaging during follow-up without new symptoms (asymptomaticRN).

At the same time, in some patients, it can give rise to new symptoms like headaches, weakness, seizures,etc (symptomatic RN). The standard treatment of RN includes steroid medicines called dexamethasone, which is helpful in a proportion of patients.

This is a prospective phase 2 study. This study is being conducted to investigate the ability of the drug Chlorophyllin in the treatment of radionecrosis.

Chlorophyllin is a water-soluble compound obtained from the green plant pigment called chlorophyll. It has been shown to have anti-cancer, anti-bacterial, anti-viral, anti-inflammatory, and antioxidant properties. It is also used as an oral formulation and is an over-the-counter drug in various countries, and also as a food colouring agent.

This is the first time chlorophyllin will be used in the setting of brain radionecrosis. Our primary aim of the study is to assess whether CHL will improve the clinical-radiological response rates. This study will be conducted on a population of 118 patients for a duration of 3 months. The total study duration is 2 years.

The study is funded by Bhabha Atomic Research Centre (BARC).

DETAILED DESCRIPTION:
Radiotherapy (RT) forms an integral role in the multi modality management of diffuse gliomas. Radiation is indicated in low-grade gliomas with high-risk features or high-grade gliomas following maximal safe resection. Higher doses of RT can lead to symptomatic radio-necrosis (RN) in approximately 5-15% of patients, typically within the first 2-3 years of RT completion. Development of RN can lead to significant morbidity with new-onset or worsening of pre-existing neurodeficit with substantial implications on quality of life, and in extreme situations, can lead to mortality as well. The pathogenesis of RN is multi factorial, with a complex interplay of vascular-mediated damage and injury to glial cells primarily postulated through the activation of several inflammatory markers like tumor necrosis factor, interleukins, and vascular endothelial growth factor. Corticosteroids, preferably dexamethasone, form the first line of management of RN, with variable response rates ranging from 25-60%, impacted by several factors like a dose of RT and response evaluation methods (neurological/ radiographic). The response rate in our practice concurs with the reported literature with combined clinical and radiological responses seen in approximately 50% of patients from institutional experience and audit. It is important to note the long-standing use of corticosteroids comes at the cost of complications like hyperglycemia, myopathy, and increased risk of infections precluding prolonged use. Also, a proportion of patients remain refractory to steroids or turn out to be dependent on steroids, where bevacizumab (anti-angiogenic agent) can be used as second-line therapy in appropriately selected patients. However, the major disadvantages of bevacizumab remain intravenous administration requiring regular hospital visits, treatment costs, and concerns for related toxicities like hypertension, and intracranial or extracranial haemorrhage. Other agents like hyperbaric oxygen therapy, pentoxifylline, and tocopherol have been suggested in refractory radionecrosis, with questionable benefits. Sodium-copper-Chlorophyllin is a phytopharmaceutical drug obtained from the green plant pigment chlorophyll. It is a semi-synthetic mixture of sodium copper salts derived from chlorophyll. Chlorophyllin scavenges RT-induced free radicals and reactive oxygen species. It is used as a food colorant and over-the-counter in the USA, Japan, Australia, and China for many years for a variety of health benefits, including prevention of body odor in geriatric patients, enhanced wound healing, antibacterial action, prevention of cancer in the high-risk population exposed to hepatocarcinogen aflatoxin B1, treatment of fecal incontinence, etc. Studies have shown that Chlorophyllin has immunostimulatory, anti-inflammatory, and antiviral effects in addition to antioxidant and radioprotective properties. It increases the expression of a transcription factor (protein) Nrf2, improving lymphocyte survival and enabling efficient detoxification after RT exposure. Chlorophyllin also delays microtubule polymerization and slows cell division in normal cells.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of diffuse glioma.
* Radionecrosis on imaging with new neurological symptoms/ worsening of prior deficits (Stratum A) or
* without new symptoms (Stratum B).
* Karnofsky Performance Scale (KPS) ≥ 50.

Exclusion Criteria:

* No tissue diagnosis.
* KPS< 50.
* Disease progression
* Contraindications to corticosteroids.
* Altered mental status with deficits in understanding or inability to consent to the study.
* Brainstem glioma
* Indeterminate for radionecrosis vs disease progression
* Prior treatment with bevacizumab (either for disease progression or radionecrosis)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Response rates | 1 month post treatment with chlorophyllin
  Clinical-radiological

SECONDARY OUTCOMES:
Survival Analysis | 3 months
  Progression-Free Survival and Overall Survival using Kaplan-Meier survival plot.
Health Questionnaire | 3 months
  EORTC QOL C -30 and (Brain module) BN-20 questionnaire. The global score and scores of subdomains will be calculated and compared with baseline.
Response rates | 3 months
  Radiological response rates at 3 months using Response Assessment in Neuro-Oncology (RANO) criteria.

OTHER OUTCOMES:
Biological response rate | 3 months
  Using functional imaging (PET & MRI) to describe the difference of SUV maximum (Maximum Standardized Uptake Value)or T/W ratio for PET scan and perfusion values e.g., rCBV ( relative Cerebral Blood Volume) for MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Archya Dasgupta, MD, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dasgupta A, Sawant S, Chatterjee A, Gota V, Sahu A, Choudhari A, Bhattacharya K, Puranik A, Dev I, Moiyadi A, Shetty P, Singh V, Menon N, Epari S, Sahay A, Shah A, Bano N, Shaikh F, Jirage A, Gupta T. Study Protocol of a Prospective Phase 2 Study of Chlorophyllin for the Management of Brain Radionecrosis in Patients With Diffuse Glioma (CHROME). Cancer Med. 2025 Mar;14(5):e70657. doi: 10.1002/cam4.70657. PMID 40025673